CLINICAL TRIAL: NCT01918397
Title: Prospective, Randomized, Blinded Phase II Pharmacokinetic/Pharmacodynamic Study of the Efficacy and Tolerability of Levofloxacin in Combination With Optimized Background Regimen for the Treatment of MDR-TB
Brief Title: Efficacy and Safety of Levofloxacin for the Treatment of MDR-TB
Acronym: Opti-Q
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency); Macleods Pharmaceuticals Ltd (Industry)
Responsible Party: Principal Investigator, Charles R Horsburgh, Professor, Epidemiology, Boston University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-32150; 1U01AI100805-01A1 (NIH)
Record Dates: First submitted 2013-08-05; First posted 2013-08-07 (Estimated); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Tuberculosis, Multidrug-Resistant
Keywords: Levofloxacin; Optimized background regimen
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — Levofloxacin; Ofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose 1 (Active Comparator): Levofloxacin 11mg/kg daily + Optimized Background Regimen (OBR)
  Interventions: Drug: Levofloxacin; Drug: Optimized background regimen (OBR)
- Dose 2 (Experimental): Levofloxacin 14mg/kg daily + Optimized Background Regimen (OBR)
  Interventions: Drug: Levofloxacin; Drug: Optimized background regimen (OBR)
- Dose 3 (Experimental): Levofloxacin 17mg/kg daily + Optimized Background Regimen (OBR)
  Interventions: Drug: Levofloxacin; Drug: Optimized background regimen (OBR)
- Dose 4 (Experimental): Levofloxacin 20mg/kg daily + Optimized Background Regimen (OBR)
  Interventions: Drug: Levofloxacin; Drug: Optimized background regimen (OBR)

INTERVENTIONS:
Drug: Levofloxacin — Levofloxacin is a quinolone antibiotic used to treat lung, sinus, skin, and urinary tract infections caused by bacteria. The chemical name is (-)-(S)-9fluoro-2,3-dihydro-3-methyl-10-(4-methyl-1-piperazinyl)-7-oxo-7H-pyrido[1,2,3-de]-1,4benzoxazine-6-carboxylic acid hemihydrate.
  Other Names: Levaquin, Quixin, and Iquix
Drug: Optimized background regimen (OBR) — For this study "OBR" will mean optimized background regimen, not including a quinolone. OBR will be selected at the discretion of the study investigator to conform with standards of care and local site guidelines. In general, the OBR regimen should include at least 3 drugs (other than levofloxacin) to which the patient's isolate is not expected to be resistant, with one of these being an injectable agent, at the usual recommended doses.

SUMMARY:
Multi-drug-resistant tuberculosis (MDR-TB) affects nearly 600,000 persons each year around the world. This type of tuberculosis is very difficult to treat, and many patients die from it. Drugs of the fluoroquinolone class are very important for treating MDR-TB, but the best dose of one of the most effective fluoroquinolones, levofloxacin, is not known. This application proposes a study to determine the best dose of levofloxacin to use in treating MDR-TB. 120 patients will receive their usual treatment, plus levofloxacin at one of four doses. The study will be performed in Peru and in South Africa, where MDR-TB is common.

DETAILED DESCRIPTION:
MDR-TB is a growing threat to international health. A recent report from WHO estimated that over 440,000 new cases of MDR-TB occurred in 127 countries in 2008, causing 150,000 deaths; this represents a 55% increase in the number of cases since 2000. Current treatment regimens have only a 58-67% success rate, and as many as 20% of those who fail to respond to treatment die of tuberculosis; those who do not die become chronic carriers and spread MDR-TB to others.

Fluoroquinolones (FQ) are an essential part of regimens for the treatment of MDR-TB; substantially better outcomes have consistently been seen in patients with MDR-TB who are treated with FQ, and newer FQ (levofloxacin, gatifloxacin and moxifloxacin) are the most potent antituberculosis agents available for MDR-TB treatment. However, gatifloxacin has been taken off the market because of dysglycemic reactions and moxifloxacin produces marked QT prolongation, increasing risk of fatal arrhythmia. In contrast, QT studies of levofloxacin have found minimal prolongation at doses up to 20mg/kg. Levofloxacin is currently given for TB at doses of 11-14 mg/kg/day and has been well tolerated at doses up to 20 mg/kg. Although the efficacy of levofloxacin increases as exposure increases both in animal studies of TB and in human studies of gram-negative bacteria, its efficacy at higher doses against TB in humans has not been studied. Thus, determination of the most efficacious and well-tolerated dose of levofloxacin is an important research priority. In this Phase 2 study, we will determine the levofloxacin dose and exposure that achieve the greatest reduction in mycobacterial burden with acceptable tolerability by studying 120 adults with smear- and culture-positive pulmonary MDR-TB at sites in Peru and South Africa. Levofloxacin will be administered with an optimized background regimen (OBR) to address the following Specific

Aims:

Specific Aim 1: To determine the levofloxacin AUC/MIC that provides the shortest time to sputum culture conversion in solid medium.

Specific Aim 2: To determine the highest levofloxacin AUC that is both safe and associated with fewer than 25% of patients discontinuing or reducing their dose of levofloxacin.

Specific Aim 3: To develop a dosing algorithm to achieve the levofloxacin AUC associated with maximal efficacy and acceptable safety/tolerability.

This clinical trial will increase our ability to cure MDR-TB and prevent the emergence of resistance to new TB drug classes by optimizing dosing and improving the effectiveness of an existing antimycobacterial agent, using a novel and versatile study design which more rapidly and efficiently identifies advances in this critical area. Construction of an algorithm to predict the optimal levofloxacin dose will allow more effective use of levofloxacin, particularly in areas with limited resources, where the burden of MDR-TB is the greatest.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with smear-positive, culture positive* pulmonary TB
2. Sputum contains isoniazid* and rifampin-resistant, Ofloxacin-susceptible MTB, all by MTBDR-sl
3. Previously treated or newly diagnosed with tuberculosis
4. Willingness to have HIV testing performed, if HIV serostatus is not known or if the last documented negative HIV test was more than 3 months prior to enrollment.
5. Age ≥ 18 years.
6. Weight > 40 Kg
7. Karnofsky score of > 60 (see section 18.1)
8. Willingness by the patient to attend scheduled follow-up visits and undergo study assessments.
9. Women with child-bearing potential must agree to use birth control if you are having sex with men while participating in this study and for three months afterward.
10. Laboratory parameters (performed within 14 days prior to enrollment):

    * Estimated Serum creatinine clearance should be <50, using nomogram78
    * Hemoglobin concentration ≥ 9.0 g/dL
    * Platelet count of ≥ 80,000/mm3
    * Absolute neutrophil count (ANC) > 1000/ mm3
    * Negative pregnancy test (for women of childbearing potential) within 14 days of enrollment
    * HIV viral load and CD4 count if HIV infected (within 3 months)
    * Serum ALT and total bilirubin <3 times upper limit of normal
11. Able to provide informed consent

Note: *Subjects may be enrolled on the basis of a presumption that they will be culture positive at either screening or baseline if they are smear-positive, but they will be excluded from the analysis if cultures are subsequently negative. This will not be deemed a protocol violation. Similarly, subjects with rifampin susceptibility on a DNA-based test may be enrolled on the basis of a presumption that they will also be INH-resistant, but they will be excluded from the analysis if the isolate is subsequently shown to be INH-susceptible. This will also not be deemed a protocol violation.

Exclusion Criteria:

1. Currently breast-feeding or pregnant.
2. Known allergy or intolerance to or toxicity from fluoroquinolones or other medications utilized in this study.
3. In the judgment of the physician the patient is not expected to survive for 6 months
4. Anticipated surgical intervention for the treatment of pulmonary tuberculosis
5. Participation in another investigational drug trial within the past 30 days
6. Concurrent use of known QT-prolonging drugs: a list of such medications can be found at http://www.azcert.org/medical-pros/drug-lists/printable-drug-list.cfm
7. Poorly controlled diabetes
8. Known g-6-phosphate dehydrogenase deficiency
9. Use of quinolone for 7 days within past 30 days
10. QTc interval greater than 450 msec for men or greater than 470 msec for women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Horsburgh, MD, Principal Investigator — Boston University
Locations (3):
- Peru (2):
  - Partners in Health, Lima
  - University of Cayetana Heredia, Lima
- Stellenbosch University, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phillips PPJ, Peloquin CA, Sterling TR, Kaur P, Diacon AH, Gotuzzo E, Benator D, Warren RM, Sikes D, Lecca L, Gandhi NR, Streicher EM, Dianis N, Eisenach K, Mitnick CD, Horsburgh CR Jr. Efficacy and Safety of Higher Doses of Levofloxacin for Multidrug-resistant Tuberculosis: A Randomized, Placebo-controlled Phase II Clinical Trial. Am J Respir Crit Care Med. 2025 Jul;211(7):1277-1287. doi: 10.1164/rccm.202407-1354OC. PMID 40080768
- [Derived] Schwalb A, Cachay R, Wright A, Phillips PPJ, Kaur P, Diacon AH, Ugarte-Gil C, Mitnick CD, Sterling TR, Gotuzzo E, Horsburgh CR. Factors associated with screening failure and study withdrawal in multidrug-resistant TB. Int J Tuberc Lung Dis. 2022 Sep 1;26(9):820-825. doi: 10.5588/ijtld.21.0729. PMID 35996282
- [Derived] van den Elsen SHJ, Sturkenboom MGG, Van't Boveneind-Vrubleuskaya N, Skrahina A, van der Werf TS, Heysell SK, Mpagama S, Migliori GB, Peloquin CA, Touw DJ, Alffenaar JC. Population Pharmacokinetic Model and Limited Sampling Strategies for Personalized Dosing of Levofloxacin in Tuberculosis Patients. Antimicrob Agents Chemother. 2018 Nov 26;62(12):e01092-18. doi: 10.1128/AAC.01092-18. Print 2018 Dec. PMID 30373800
- [Derived] Peloquin CA, Phillips PPJ, Mitnick CD, Eisenach K, Patientia RF, Lecca L, Gotuzzo E, Gandhi NR, Butler D, Diacon AH, Martel B, Santillan J, Hunt KR, Vargas D, von Groote-Bidlingmaier F, Seas C, Dianis N, Moreno-Martinez A, Kaur P, Horsburgh CR Jr. Increased Doses Lead to Higher Drug Exposures of Levofloxacin for Treatment of Tuberculosis. Antimicrob Agents Chemother. 2018 Sep 24;62(10):e00770-18. doi: 10.1128/AAC.00770-18. Print 2018 Oct. PMID 30012767
- [Derived] Bouton TC, Phillips PPJ, Mitnick CD, Peloquin CA, Eisenach K, Patientia RF, Lecca L, Gotuzzo E, Gandhi NR, Butler D, Diacon AH, Martel B, Santillan J, Hunt KR, Vargas D, von Groote-Bidlingmaier F, Seas C, Dianis N, Moreno-Martinez A, Horsburgh CR Jr. An optimized background regimen design to evaluate the contribution of levofloxacin to multidrug-resistant tuberculosis treatment regimens: study protocol for a randomized controlled trial. Trials. 2017 Nov 25;18(1):563. doi: 10.1186/s13063-017-2292-x. PMID 29178937

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4
Started | 27 | 29 | 28 | 27
Completed | 16 | 21 | 20 | 20
Not Completed | 11 | 8 | 8 | 7
Not completed — Never started treatment | 2 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 0
Not completed — Lack of compliance | 2 | 2 | 3 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Rifampin susceptible | 0 | 0 | 0 | 2
Not completed — Treatment failure | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 1 | 1
Not completed — XDR at baseline | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1 | 1
Not completed — Increased QTc | 1 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Involved in another investigative trial | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Total
Number analyzed (Participants) | 27 | 29 | 28 | 27 | 111
Age, Customized [Median (Inter-Quartile Range); unit: years] | 32 [25 to 43] | 25 [23 to 31] | 26 [22 to 37.5] | 31 [21 to 44] | 26 [22 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 10 | 14 | 43
  Male | 17 | 20 | 18 | 13 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 17 | 16 | 15 | 62
  Not Hispanic or Latino | 12 | 12 | 12 | 12 | 48
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 5 | 7 | 6 | 6 | 24
  Other | 22 | 22 | 22 | 21 | 87
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 12 | 12 | 12 | 12 | 48
  Peru | 15 | 17 | 16 | 15 | 63

OUTCOME MEASURES:

1. Primary Outcome: Time to Sputum Culture Conversion
Description: The primary efficacy endpoint is the time to sputum culture conversion from positive to negative for M. tuberculosis growth on solid medium. This is defined as the time from initiation of study treatment to the first of two successive negative cultures one study visit apart that are not followed by a culture-positive specimen within 28 weeks of treatment initiation. To ensure that each subject will be evaluable for the primary endpoint, bi-weekly sputum cultures will be collected for 12 weeks, then every 4 weeks through 24 weeks of treatment.
Time Frame: 28 weeks
Population: A modified intention to treat (MITT) population n=98 was analyzed.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4
Number analyzed (Participants) | 24 | 27 | 24 | 23
weeks | 5.9 [2.3 to 10.1] | 6.3 [4.1 to 10.0] | 6.1 [4.1 to 10.1] | 6.1 [4.0 to 8.1]

2. Primary Outcome: Number of Grade 3,4, and 5 AEs
Description: The primary safety endpoint will be the number of grade 3, 4 and 5 adverse events (AEs), occurring up to and including the time on study drug plus four weeks post study drug completion.
Time Frame: 28 weeks
Population: Intention to treat analysis based on the number of participants that completed treatment (n=108).
Measure: Number; unit: Events
Units Other Than Participants: Events
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4
Number analyzed (Participants) | 25 | 28 | 28 | 27
Number analyzed (Events) | 421 | 419 | 461 | 519
Events | 5 | 4 | 14 | 13

3. Secondary Outcome: Number of Patients Completing Treatment
Description: The primary endpoint for the analysis of tolerability will be the ability to complete 24 weeks of treatment with the assigned levofloxacin dose (in mg/kg at enrollment).
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4
Number analyzed (Participants) | 25 | 28 | 28 | 27
Participants | 23 | 26 | 27 | 24

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signing of consent form to the final visit. For a typical participant that would be 28 weeks.
Description: The definitions do not differ from the clinicaltrials.gov definitions.
Arm/Group | Dose 1 | Dose 2 | Dose 3 | Dose 4
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/28 | 1/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 2/25 | 1/28 | 4/28 | 3/27
Other Adverse Events (participants affected / at risk) | 24/25 | 28/28 | 28/28 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 (N=25) | Dose 2 (N=28) | Dose 3 (N=28) | Dose 4 (N=27)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremily (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose 1 (N=25) | Dose 2 (N=28) | Dose 3 (N=28) | Dose 4 (N=27)
Blood uric acid increased (Investigations) | 2 | 5 | 2 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Deafness (Ear and labyrinth disorders) | 3 | 3 | 5 | 3
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 3 | 6 | 5 | 4
Decreased appetite (Metabolism and nutrition disorders) | 5 | 4 | 4 | 12
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 16 | 13 | 13 | 17
Drug induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Meningitis Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 | 11 | 16 | 17
Nausea (Gastrointestinal disorders) | 17 | 14 | 19 | 20
Neuropathy peripheral (Nervous system disorders) | 1 | 3 | 4 | 4
Oedema peripheral (General disorders) | 0 | 1 | 2 | 3
Ototoxicity (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 4 | 3 | 5 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 11 | 15 | 8 | 15
Acariasis (Infections and infestations) | 0 | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 2
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Affect Lability (Psychiatric disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 3 | 0
Anorectal disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 5
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 19 | 18 | 22
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Aspartate Aminostransferase Increased (Investigations) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 4 | 3
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 1 | 0
Blood folate decreased (Investigations) | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1
Body Tinia (Infections and infestations) | 0 | 2 | 0 | 0
Bradycardia (Cardiac disorders) | 4 | 4 | 4 | 6
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 1 | 1
Breath sounds abnormal (Investigations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Bulimia Nervosa (Psychiatric disorders) | 0 | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Conjunctivitis Allergic (Eye disorders) | 0 | 0 | 1 | 1
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 6 | 4 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 0
costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 4 | 2
Creatinine Renal Clearance (Investigations) | 0 | 2 | 1 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dental Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 2
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1
Diabetes Mellitus (Endocrine disorders) | 1 | 0 | 0 | 0
Diarrrhoea (Gastrointestinal disorders) | 6 | 6 | 8 | 10
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 5 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 3 | 2 | 0
Ear Discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 3 | 3 | 3
Eosinophil Count Increase (Investigations) | 1 | 0 | 0 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Exoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Eye Pruritis (Eye disorders) | 0 | 0 | 1 | 1
Eye Swelling (Eye disorders) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 2
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Fungal Infection (Infections and infestations) | 1 | 1 | 2 | 0
Gastric Disorder (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 5 | 5 | 5 | 9
Gastroenteritis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gastrooesophageal reflux (Gastrointestinal disorders) | 2 | 1 | 1 | 3
Gingival Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Grip strength decreased (Investigations) | 0 | 1 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 5 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Hallucinations, mixed (Psychiatric disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 11 | 13 | 13 | 13
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 2 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2 | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 4 | 3 | 5
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 2 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 8 | 2 | 2 | 7
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 3 | 0 | 0 | 3
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 7 | 7 | 3 | 6
Insomnia (Psychiatric disorders) | 10 | 6 | 6 | 8
Jaundice (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 2
Libido increased (Psychiatric disorders) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 1 | 2
Mood altered (Psychiatric disorders) | 0 | 1 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 3
Myopia (Eye disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 4 | 1 | 3
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neuritis (Nervous system disorders) | 1 | 0 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 3
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Oral Candidiasis (Infections and infestations) | 1 | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Otitis Externa (Infections and infestations) | 0 | 1 | 0 | 1
Otitis Media (Infections and infestations) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 6 | 7 | 9
Pallor (Vascular disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 2 | 7 | 2 | 5
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 3 | 1 | 0 | 3
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Personality disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 4 | 0
Pharyngitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Physical assault (Social circumstances) | 0 | 0 | 0 | 1
Pityriasis alba (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 2 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Post herpetic Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Post inflammatory pigment change (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 13 | 18 | 13
Pruritus genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Psoas Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 3 | 0 | 0
Pyrexia (General disorders) | 5 | 7 | 3 | 4
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 8 | 9 | 14 | 15
Rash pustular (Infections and infestations) | 0 | 1 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 2 | 5 | 4
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Transaminases increased (Investigations) | 0 | 0 | 2 | 1
Tremor (Nervous system disorders) | 2 | 1 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 2 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 2
Vessel puncture site bruise (General disorders) | 0 | 1 | 1 | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 2 | 3
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 13 | 14 | 15 | 15
Vulvovaginitis (Infections and infestations) | 0 | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Xerosis (General disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT01918397/Prot_SAP_000.pdf